CLINICAL TRIAL: NCT05028322
Title: Effectiveness and Safety of Intra-Dermal Hepatitis B Vaccination After Topical Application of IMIQUIMOD, in Cirrhotics Patients, Who Did Not Respond to the Conventional Vaccine Regimen: a Pilot Study
Brief Title: Evaluation of Intradermal Hepatitis B Vaccine After IMIQUIMOD's Application, in Cirrhotics Who Did Not Respond to the Usual Vaccine Regimen
Acronym: IDMODVHB
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021-000644-22
Record Dates: First submitted 2021-07-06; First posted 2021-08-31 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-06

CONDITIONS: Cirrhosis, Liver; Vaccination Failure; HBV; Vaccine Reaction
MeSH Terms: conditions — Liver Cirrhosis | interventions — Hepatitis B Surface Antigens

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intra-muscular vaccination (Group 1) (Active Comparator): This group corresponds to the use of the vaccine as used in the current recommendations.
  Interventions: Biological: HEPATITIS B SURFACE ANTIGEN
- Intra-dermal vaccination group without application of IMIQUIMOD cream (Group 2) (Active Comparator): Administration mode change for Intra-dermal vaccination. ( Instead of Intra-musculaire ) , to have a comparative with the experimental group.
  Interventions: Biological: HEPATITIS B SURFACE ANTIGEN
- Intra-dermal vaccination group with application of IMIQUIMOD cream (Group 3) (Experimental): Intra-dermal vaccin administration, with an immunity booster few minutes before by IMIQUIMOD application cream.
  Experimental group.
  Interventions: Drug: IMIQUIMOD cream; Biological: HEPATITIS B SURFACE ANTIGEN

INTERVENTIONS:
Drug: IMIQUIMOD cream — Cream to apply before intra-dermal vaccine injection
  Arms: Intra-dermal vaccination group with application of IMIQUIMOD cream (Group 3)
Biological: HEPATITIS B SURFACE ANTIGEN — HBV Vaccine

SUMMARY:
In a population of cirrhotics patients who did not responde to an anti-HBV vaccination according to the recommended vaccination, the goal is to :

Describe the proportion of patients with HBs antibody levels greater than 10mUI/mL at 1 month of the last injection of vaccine ; with a M0-M1-M6 vaccine regimen using 3 vaccines strategies :

* After simple intramuscular vaccine (IM) ( Control group )
* After simple intradermal vaccine
* after IMIQUIMOD's application followed by intradermal vaccine administration

The main hypothesis of this study is : IMIQUIMOD acts as an immunity booster, so the combination of IMIQUIMOD with an intra-dermal injection of the anti-HBV vaccine allows better acquisition of post-vaccination immunization.

DETAILED DESCRIPTION:
This study will be in a population of Cirrhotic patients who have already received a HBV vaccination with a conventional regimen and who have not responded (characterized by a level of antibody Hbs < 10UI/ml at the end of the vaccine regimen).

In current recommendations, up to 3 additional injections of HBV vaccine should be injected to obtain an antibody level> 10 mIU / ml.

In this study, the investigator will describe the proportion of patients with HBs antibody levels greater than 10mUI/mL at 1 month of the last injection of vaccine ; with a M0-M1-M6 vaccine regimen using 3 vaccines strategies :

* After simple intramuscular vaccine (IM) ( Control group )
* After simple intradermal vaccine
* after IMIQUIMOD's application followed by intradermal vaccine administration

ELIGIBILITY:
Inclusion Criteria:

* Adults (> 18 years old)

  * Cirrhotic patient, all etiologies except related to chronic HBV infection.
  * Cirrhotic patient who did not respond to a 1st conventional hepatitis B vaccination regimen administered intramuscularly (ac Anti HBs < 10 mUI/ml)
  * Person affiliated to a social security plan
  * Person who received complete information about the organization of the research and who signed informed consent

Exclusion Criteria:

* Patients with contraindication to the use of an intramuscular vaccine : Patients on Anticoagulants; Hemophiliac Patients, Patients with Severe Hemostasis Disorder (objectified by TP < 30%; and/or a Thombopenia with platelets < 30G/L)
* Patients with end-stage chronic kidney failure defined by DFG <15ml/min/1.73m2 _ Hemodialysised Patients
* Patients with a skin condition that does not allow vaccination (intradermal or intra-muscle): Skin sores on both arms: ulcers/abrasions/bubbles ; without healthy skin intervals.
* Femme of childbearing age who does not have an effective method of contraception for the duration of the study. Effective contraceptive methods are defined as combined hormonal contraception (containing estrogen and progestin) combined with ovulation inhibition (oral, intravaginal, transdermal); or progestin-only hormonal contraception combined with ovulation inhibition (oral, injectable, implantable); or intrauterine device (IUD); or intrauterine hormone delivery system (IUS); or bilateral tubal occlusion; or a vasectomized partner; or sexual abstinence; Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. Menopause is defined as the absence of menstruation for at least 12 months. According to CTFG recommendations related to contraception and pregnancy testing in clinical trials; version 1.1 of 21/09/2020.
* Personne referred to sections L. 1121-5, L. 1121-7 and L1121-8 of the Public Health Code. Pregnant, parturient or breastfeeding mother Minor (unassecipated) An adult subject to a legal protection measure (tutelage, curate, safeguarding of justice) Adult person undying to express consent
* Persons deprived of liberty by judicial or administrative decision, persons receiving psychiatric care under sections L. 3212-1 and L. 32131.
* Vaccination during the 4 weeks (28 days) prior to the first vaccination in the trial
* Previous vaccination with another investigational vaccine
* Subjects who have received immunoglobulins, blood or blood derivatives within the last 3 months.
* Known or suspected congenital or acquired immunodeficiency; immunosuppressive therapy within the last 6 months, such as cancer chemotherapy or radiotherapy; long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the last 3 months).
* Acute respiratory infection or severe acute febrile illness (temperature ≥ 38.0°C), or a systemic reaction that may be of significant risk with vaccination in the month prior to inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients in each groups, with HBs antibody levels greater than 10mUI/mL at 1 month of the last injection of vaccine | 1 month of the last injection of vaccine, it means 1 month after the end of the total procedure.
  Describe the proportion of patients with HBs antibody levels greater than 10mUI/mL at 1 month of the last injection of vaccine ; with a M0M1-M6 vaccine regimen using 3 vaccines strategies:
  * After simple intramuscular vaccine (IM) ( Control group , group 1)
  * After simple intradermal vaccine without IMIQUIMOD ( Group 2 )
  * after IMIQUIMOD's application followed by intradermal vaccine administration ( Group 3 )

SECONDARY OUTCOMES:
Describe the proportion of patients with an anti-HB antibody level greater than 10mUI/mL at 1 month of the first injection (M1) with a vaccine regimen according to the vaccine strategy | 1 month of the first vaccine injection (Month 1)
  Rate of patients with an anti-HB antibody level greater than 10mUI/mL at 1 month of the first injection (M1) with a vaccine regimen according to the vaccine strategy
Describe the proportion of patients with an anti-HB antibody level greater than 10mUI/mL at 6 months of the first injection (M6) with a vaccine regimen according to the vaccine strategy | 6 months of the first vaccine injection (Month 6)
  Rate of patients with an anti-HB antibody level greater than 10mUI/mL at 6 months of the first injection (M6) with a vaccine regimen according to the vaccine strategy
Describe the evolution of the level of anti-HBs antibodies between 2 successive visits according to the vaccine strategy | -Day 0 / Month 0 ; - Day 30 / Month 1 ; - Day 180 / Month 6 ; - Day 210 / Month 7
  * Anti-HBs Antibodies Level in the first vaccine injection = Day 0 / Month 0
  * Antibodies Level in the second vaccine injection = 30 days (1 month) after the first injection.
  * Antibodies Level in the third vaccine injection = 180 days (6months) after the first vaccine injection (or 150 days/5months after the second vaccine injection)
  * Antibodies Level at the end of the study : 210 days (7 months) after the first injection ; (or 30 days/1month after the third injection ) ;
Describe the rate of adverse events (by severity level) following the injection of a dose of intradermal vaccine | In each visit ( Month 1 , Month 6 , Month 7 )
  In each visit ( Month 1 , Month 6 , Month 7 ) we describe the rate of adverse events (by severity level) following the injection of a dose of intradermal vaccine
Describe the rate of adverse events (by severity level) following the injection of an intradermal vaccine dose after prior application of Imiquimod | In each visit ( Month 1 , Month 6 , Month 7 )
  In each visit ( Month 1 , Month 6 , Month 7 ) we describe the rate of adverse events (by severity level) after injection of an intradermal vaccine dose after prior application of Imiquimod